CLINICAL TRIAL: NCT01255930
Title: Evaluation of Placenta Maturity by the Sonographic Textures
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Szu-Yuan Chou, Obsterics & Gynecology
Other Study IDs: 99016
Record Dates: First submitted 2010-12-06; First posted 2010-12-08 (Estimated); Last update posted 2010-12-08 (Estimated); Status verified 2010-12

CONDITIONS: Pregnant Women
Keywords: Pregnant Women; Sonographic Textures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to evaluate placenta maturity by the sonographic textures.The evaluation of placenta maturity by the sonographic textures is related to anticipative pregnancy and actual pregnancy . By analyzing this theory, the investigators want to bring up another objective and accurate analysis method in order to provide information for the evaluation of clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women
* Placenta Maturity by the Sonographic Textures

Exclusion Criteria:

* intrauterine-growth retardation(IUGR)
* Pre-eclampsia
* Higher Blood Pressure
* Fetal Distress during a labor

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: pregnant women
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2010-01; Study Completion 2011-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Szu-Yuan Chou, Principal Investigator — Taipei Medical University WanFang Hospital
Locations (1):
- Taipei Medical University-WanFang Hospital, Taipei, Taiwan